CLINICAL TRIAL: NCT06467357
Title: DESTINY-Biliary Tract Cancer-01: A Phase 3 Study of Trastuzumab Deruxtecan (T-DXd) and Rilvegostomig Versus Standard-of-Care Gemcitabine, Cisplatin, and Durvalumab for First Line Locally Advanced or Metastatic HER2-expressing Biliary Tract Cancer
Brief Title: Phase 3 Study of T-DXd and Rilvegostomig Versus SoC in Advanced HER2-expressing Biliary Tract Cancer
Acronym: DESTINY-BTC01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D781PC00001; 2023-508057-19-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-05-21; First posted 2024-06-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; HER2; HER2 expressing BTC; Trastuzumab deruxtecan; T-DXd; Rilvegostomig
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; durvalumab; trastuzumab deruxtecan

STUDY DESIGN:
Masking Description: This is an open-label, Sponsor-blinded study. To maintain the integrity of the study, Sponsor personnel directly involved in study conduct will not undertake or have access to efficacy data aggregated by treatment group prior to final data readout for the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trastuzumab deruxtecan + rilvegostomig (Experimental): Trastuzumab deruxtecan (T-DXd; DS-8201a) in combination with rilvegostomig arm
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Rilvegostomig
- Trastuzumab deruxtecan (Experimental): Trastuzumab deruxtecan (T-DXd; DS-8201a) arm
  Interventions: Drug: Trastuzumab deruxtecan
- Standard of Care (Active Comparator): Gemcitabine and cisplatin in combination with durvalumab arm
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab

INTERVENTIONS:
Drug: Gemcitabine — Standard of care chemotherapy by intravenous infusion
  Arms: Standard of Care
Drug: Cisplatin — Standard of care chemotherapy by intravenous infusion
  Arms: Standard of Care
Drug: Durvalumab — Standard of care immunotherapy by intravenous infusion
  Arms: Standard of Care
Drug: Trastuzumab deruxtecan — Experimental therapy by intravenous infusion
  Other Names: DS-8201a; T-DXd
  Arms: Trastuzumab deruxtecan; Trastuzumab deruxtecan + rilvegostomig
Drug: Rilvegostomig — Experimental therapy by intravenous infusion
  Arms: Trastuzumab deruxtecan + rilvegostomig

SUMMARY:
The purpose of this study is to measure the efficacy and safety of T-DXd with rilvegostomig or T-DXd monotherapy compared with gemcitabine plus cisplatin and durvalumab in patients with advanced treatment naïve HER2-expressing BTC.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients must be at least 18 years of age at the time of signing the informed consent. Other age restrictions may apply as per local regulations.
* Unresectable, previously untreated, locally advanced or metastatic biliary tract adenocarcinoma. Prior treatment in the perioperative and/or adjuvant setting is permissible provided there is > 3 months (90 days) between the end of adjuvant treatment and the diagnosis of locally advanced or metastatic disease.
* Histologically confirmed HER2-expressing (IHC 3+ or IHC 2+) BTC.
* Patients must provide an FFPE tumor sample that is no older than 3 years for tissue-based IHC staining to centrally determine HER2 expression, PD-L1 status, and other correlatives.
* Has at least one target lesion assessed by the Investigator based on RECIST v1.1. (Randomized portion only)
* WHO/ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
* Adequate organ and bone marrow function within 14 days before randomization.
* Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential.
* Minimum life expectancy of 12 weeks.

Key Exclusion Criteria:

* Prior exposure to other HER2 targeting therapies, ADCs, immune checkpoint inhibitors and therapeutic anticancer vaccines.
* Histologically confirmed ampullary carcinoma.
* Any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the Investigator, interfere with the patient's participation in the clinical study or evaluation of the clinical study results.
* Spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Medical history of myocardial infarction within 6 months before randomization/enrollment, symptomatic congestive heart failure (New York Heart Association Class II to IV), unstable angina pectoris, clinically important cardiac arrhythmias, or a recent (< 6 months) cardiovascular event including stroke.
* Serious chronic gastrointestinal conditions associated with diarrhea (eg, active inflammatory bowel disease); active non-infectious skin disease (including any grade rash, urticaria, dermatitis, ulceration, or psoriasis) requiring systemic treatment.
* Active autoimmune, connective tissue or inflammatory disorders that has required systemic treatment in the past 2 years, or where there is documented, or a suspicion of pulmonary involvement at the time of screening.
* Corrected QT interval (QTcF) prolongation to > 470 msec (females) or > 450 msec (males) based on average of the screening triplicate 12-lead ECG.
* History of (non-infectious) ILD/pneumonitis, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion etc).
* Prior pneumonectomy (complete).
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals. Patients with prior cholangitis/biliary tract infections/biliary intervention (eg, stent, external drain) should have completed a full course of antibiotics prior to randomization.
* Active primary immunodeficiency, known uncontrolled active HIV infection or HCV.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 3 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected nonmelanoma skin cancer and curatively treated in situ disease. For certain participant populations, exceptions could also include carcinomas in-situ or Ta tumors treated with curative intent.
* Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (Drainage and Cell free and Concentrated Ascites Reinfusion Therapy are not allowed within 2 weeks prior to screening assessment).
* Any concurrent anticancer treatment without an adequate washout period prior to randomization. Concurrent use of hormonal therapy for non-cancer related conditions (eg, hormone replacement therapy) is allowed.
* History of organ transplants or allogenic stem cell transplant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2028-06-12 (Estimated); Study Completion 2029-05-16 (Estimated)

PRIMARY OUTCOMES:
Safety Run In: To evaluate the safety and tolerability of T-DXd with rilvegostomig | Until all patients have completed at least 1 full Cycle (each cycle is 21 days)
  Safety and tolerability will be evaluated by the proportion of treated patients with occurrence of AEs, SAEs and AESIs, as assessed by CTCAE v5.0.
Randomized Portion: To evaluate the efficacy of T-DXd with rilvegostomig vs Standard of Care (SoC) in terms of Overall Survival in the FAS (HER2 IHC 3+) population | From date of treatment randomization until the date of death from any cause (estimated to be assessed up to 50 months after first subject randomized)
  Overall survival (OS) in FAS (HER2 IHC 3+) population OS is defined as time from randomization date until the date of death due to any cause. The comparison will include all randomized patients, regardless of whether the patient withdraws from therapy or receives another anticancer therapy. The measure of interest is the hazard ratio of OS.

SECONDARY OUTCOMES:
To evaluate the efficacy of T-DXd with rilvegostomig vs Standard of Care in terms of Overall Survival in the FAS (HER2 IHC 3+/2+) population | From date of randomization until the date of death from any cause (estimated to be assessed up to 50 months after first subject randomized)
  Overall Survival (OS) in FAS (HER2 IHC 3+/2+) population. OS definition as above.
To evaluate the efficacy of T-DXd monotherapy vs Standard of Care in terms of Overall Survival in the FAS (HER2 IHC 3+) population | From date of randomization until the date of death from any cause (estimated to be assessed up to 50 months after first subject randomized)
  Overall Survival (OS) in FAS (HER2 IHC 3+) population. OS definition as above.
To evaluate the efficacy of T-DXd monotherapy vs Standard of Care in terms of Overall Survival in the FAS (HER2 IHC 3+/2+) population | From date of randomization until the date of death from any cause (estimated to be assessed up to 50 months after first subject randomized)
  Overall Survival (OS) in FAS (HER2 IHC 3+/2+) population. OS definition as above.
To further evaluate efficacy of T-DXd with rilvegostomig vs Standard of Care in terms of Progression Free Survival in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Progression free survival (PFS) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  PFS is defined as time from randomization until progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients, regardless of whether the patient withdraws from randomized therapy, receives another anticancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the hazard ratio of PFS.
To further evaluate efficacy of T-DXd monotherapy vs Standard of Care in terms of Progression Free Survival in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Progression free survival (PFS) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  PFS is defined as time from randomization until progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients, regardless of whether the patient withdraws from randomized therapy, receives another anticancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the hazard ratio of PFS.
To further evaluate the efficacy of T-DXd with rilvegostomig vs Standrad of Care in terms of objective response rate in the FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Objective response rate (ORR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  ORR is defined as the proportion of patients who achieved CR or PR per RECIST 1.1, as assessed by the investigator. The analysis will include objective response data for all randomized patients from randomization until progression, or up to the last evaluable assessment in the absence of progression.
  Patients who go off-treatment without a response or progression and then respond while receiving a subsequent therapy will not be included as responders in the ORR calculation.
  The measure of interest is the risk difference of ORR.
To further evaluate the efficacy of T-DXd monotherapy vs Standrad of Care in terms of objective response rate in the FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Objective response rate (ORR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  ORR is defined as the proportion of patients who achieved CR or PR per RECIST 1.1, as assessed by the investigator. The analysis will include objective response data for all randomized patients from randomization until progression, or up to the last evaluable assessment in the absence of progression.
  Patients who go off-treatment without a response or progression and then respond while receiving a subsequent therapy will not be included as responders in the ORR calculation.
  The measure of interest is the risk difference of ORR.
To further evaluate efficacy of T-DXd with rilvegostomig vs Standard if Care in terms of duration of response in patients with HER2-expressing BTC in the FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From the date of first documented response until date of documented progression or death due to any cause, whichever occurs first (estimated up to 50 months)
  Duration of response (DoR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  DoR will be defined as the time from the date of first documented response until date of documented progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients who have a response, regardless of whether the patient withdraws from randomized therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the median DoR.
To further evaluate efficacy of T-DXd monotherapy vs Standard if Care in terms of duration of response in patients with HER2-expressing BTC in the FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From the date of first documented response until date of documented progression or death due to any cause, whichever occurs first (estimated up to 50 months)
  Duration of response (DoR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  DoR will be defined as the time from the date of first documented response until date of documented progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients who have a response, regardless of whether the patient withdraws from randomized therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the median DoR.
To further evaluate the efficacy of T-DXd with rilvegostomig versus T-DXd monotherapy in terms of Overall survival in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations. | From date of randomization until the date of death from any cause (estimated to be assessed up to 50 months after first subject randomized)
  Overall survival (OS) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  OS is defined as time from randomization date until the date of death due to any cause. The comparison will include all randomized patients, regardless of whether the patient withdraws from therapy or receives another anticancer therapy. The measure of interest is the hazard ratio of OS.
To further evaluate the efficacy of T-DXd with rilvegostomig versus T-DXd monotherapy in terms of PFS in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From the date of randomisation until progression or death due to any cause, whichever occurs first (estimated up to 50 months)
  Progression free survival (PFS) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  PFS is defined as time from randomization until progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients, regardless of whether the patient withdraws from randomized therapy, receives another anticancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the hazard ratio of PFS.
To further evaluate the efficacy of T-DXd with rilvegostomig versus T-DXd monotherapy in terms of Duration of response in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From the date of first response until progression or death due to any cause, whichever occurs first (estimated up to 50 months)
  Duration of response (DoR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  DoR will be defined as the time from the date of first documented response until date of documented progression per RECIST v1.1, or death due to any cause. The analysis will include all randomized patients who have a response, regardless of whether the patient withdraws from randomized therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST v1.1 progression.
  The measure of interest is the median DoR.
To further evaluate the efficacy of T-DXd with rilvegostomig versus T-DXd monotherapy in terms of Objective response rate in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Objective response rate (ORR) in FAS (HER2 IHC 3+) and FAS (HER2 IHC 3+/2+) populations.
  ORR is defined as the proportion of patients who achieved CR or PR per RECIST 1.1, as assessed by the investigator. The analysis will include objective response data for all randomized patients from randomization until progression, or up to the last evaluable assessment in the absence of progression.
  Patients who go off-treatment without a response or progression and then respond while receiving a subsequent therapy will not be included as responders in the ORR calculation.
  The measure of interest is the risk difference of ORR.
To assess the safety and tolerability of T-DXd with rilvegostomig vs Standard of Care | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Safety and tolerability will be evaluated by the proportion of treated patients with occurrence of AEs, SAEs and AESIs, as assessed by CTCAE v5.0.
To assess the safety and tolerability of T-DXd monotherapy vs Standard of Care | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Safety and tolerability will be evaluated by the proportion of treated patients with occurrence of AEs, SAEs and AESIs, as assessed by CTCAE v5.0.
To describe patient-reported tolerability of T-DXd with rilvegostomig in comparison to Standard of Care based on a summary of symptomatic AEs | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Symptomatic adverse events: Descriptive summary of the proportion of patients reporting symptomatic AEs while on treatment using items from the EORTC Item Library (on EORTC IL form 322).
To describe patient-reported tolerability of T-DXd monotherapy in comparison to SoC based on a summary of symptomatic AEs | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Symptomatic adverse events: Descriptive summary of the proportion of patients reporting symptomatic AEs while on treatment using items from the EORTC Item Library (on EORTC IL form 322)
To describe patient-reported tolerability of T-DXd with rilvegostomig in comparison to T-DXd monotherapy based on a summary of symptomatic AEs | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Symptomatic adverse events: Descriptive summary of the proportion of patients reporting symptomatic AEs while on treatment using items from the EORTC Item Library (on EORTC IL form 322).
To assess time to deterioration in physical functioning in patients treated with T-DXd with rilvegostomig vs Standard of Care | Until End of Study (estimated up to 50 months)
  Time to deterioration (TTD) in physical function as measured by the PROMIS Short Form v2.0 - Physical Function 8c - TTD is defined as time from the date of randomization to the date of deterioration.
  Deterioration is defined as the change from baseline that reaches a clinically meaningful deterioration threshold.
  - The measure of interest is the HR of TTD in physical function. The analysis will include all randomized patients as randomized.
To assess time to deterioration in physical functioning in patients treated with T-DXd monotherapy vs Standard of care | Until End of Study (estimated up to 50 months)
  Time to deterioration (TTD) in physical function as measured by the PROMIS Short Form v2.0 - Physical Function 8c - TTD is defined as time from the date of randomization to the date of deterioration.
  Deterioration is defined as the change from baseline that reaches a clinically meaningful deterioration threshold.
  - The measure of interest is the HR of TTD in physical function. The analysis will include all randomized patients as randomized.
To assess time to deterioration in physical functioning in patients treated with T-DXd with rilvegostomig vs T-DXd monotherapy | Until End of Study (estimated up to 50 months)
  Time to deterioration (TTD) in physical function as measured by the PROMIS Short Form v2.0 - Physical Function 8c - TTD is defined as time from the date of randomization to the date of deterioration.
  Deterioration is defined as the change from baseline that reaches a clinically meaningful deterioration threshold.
  - The measure of interest is the HR of TTD in physical function. The analysis will include all randomized patients as randomized.
To assess the pharmacokinetics of T-DXd, total anti- HER2 antibody, DXd and rilvegostomig in serum | From the time of informed consent until 90 days after the last dose of T-DXd and rilvegostomig
  Descriptive analysis of serum concentration of T-DXd, total anti-HER2 antibody, DXd and rilvegostomig in all applicable arms.
To investigate the immunogenicity of T-DXd and of rilvegostomig | From the time of informed consent until 30 and 90 days after the last dose of T-DXd and rilvegostomig, respectively
  Descriptive summary of presence of ADAs for T-DXd and rilvegostomig in all applicable arms.
To describe patient-reported tolerability of T-DXd with rilvegostomig in comparison to Standard of Care based on overall side-effect bother | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Overall side-effect bother that will be mesured using PGI-TT
To describe patient-reported tolerability of T-DXd monotherapy in comparison to SoC based on overall side-effect bother | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Overall side-effect bother that will be assessed will be mesured using PGI-TT
To assess the safety and tolerability of T-DXd with rilvegostomig vs T-DXd monotherapy | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first (estimated to be assessed up to 50 months)
  Safety and tolerability will be evaluated by the proportion of treated patients with occurrence of AEs, SAEs and AESIs, as assessed by CTCAE v5.0.
To describe patient-reported tolerability of T-DXd with rilvegostmog in comparison to T-DXd monotherapy based on overall side-effect bother | Until End of Study (estimated up to 50 months)
  Patient-reported tolerability will be described using the Overall side-effect bother that will be assessed will be mesured using PGI-TT.

CONTACTS AND LOCATIONS:
Locations (219):
- United States (37):
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Towson, Maryland
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, White Plains, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Australia (4):
  - Research Site, Chermside
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Nedlands
- Austria (5):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
- Belgium (6):
  - Research Site, Anderlecht
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (5):
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Santa Maria
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (30):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linyi
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (9):
  - Research Site, Brest
  - Research Site, Clichy
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Pessac
  - Research Site, Villejuif
- Germany (13):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Ulm
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (7):
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (8):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Naples
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Tricase
- Japan (26):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuyama-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kita-gun
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Suita
  - Research Site, Sunto-gun
  - Research Site, Ube-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Research Site, Rotterdam, Netherlands
- Philippines (4):
  - Research Site, Cebu City
  - Research Site, Makati
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Saudi Arabia (2):
  - Research Site, Dammam
  - Research Site, Riyadh
- Slovakia (5):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Martin
  - Research Site, Trnava
- South Korea (5):
  - Research Site, Busan
  - Research Site, Gyeonggi-do
  - Research Site, Hwasun-gun
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santander
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (8):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Mueang
  - Research Site, Naimuang
  - Research Site, Ongkharak
  - Research Site, Si Sa Ket
- Turkey (Türkiye) (6):
  - Research Site, Altındağ
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mezitli
  - Research Site, Yakutiye
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Greater London
  - Research Site, Leeds
  - Research Site, London
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home